CLINICAL TRIAL: NCT02237846
Title: Clinical Study of Umbilical Cord Tissue Mesenchymal Stem Cells (UC-MSC) for Treatment of Osteoarthritis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No enrollment
Sponsor: Translational Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNEI-2014-TBS-UCMSCOA-001
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee; stem cells; mesenchymal; umbilical cord
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intra-articular knee injection of UC-MSC (Active Comparator): Human umbilical cord tissue-derived mesenchymal stem cells administered into the knee joint once
  Interventions: Biological: Human umbilical cord tissue-derived mesenchymal stem cells
- IV injection of UC-MSC (Active Comparator): Human umbilical cord tissue-derived mesenchymal stem cells administered once per day for 3 consecutive days
  Interventions: Biological: Human umbilical cord tissue-derived mesenchymal stem cells

INTERVENTIONS:
Biological: Human umbilical cord tissue-derived mesenchymal stem cells

SUMMARY:
Allogeneic human umbilical cord tissue-derived stem cells injected intravenously (IV) once per day for 3 days or once intra-articularly are a safe and will induce a therapeutic effect in osteoarthritis (OA) patients.

DETAILED DESCRIPTION:
The proposed study will assess primarily safety and secondary efficacy endpoints of allogeneic umbilical cord mesenchymal stem cells (UC-MSC) administered to 40 patients with OA. Arm 1 will receive one intra-articular injection of UC-MSC into the knee and Arm 2 will receive IV UC-MSC once per day for 3 consecutive days.

The primary objective of the trial is freedom from treatment associated adverse events at 3 and 12 months post treatment. Secondary objective will be efficacy as assessed at baseline, and 3 and 12 months post treatment and will be quantified based on the Western Ontario and McMaster osteoarthritis index (WOMAC).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by the subject.
* Age greater than or equal to 18 years
* Ability to understand the planned treatment.
* Idiopathic or secondary osteoarthritis of the knee with grade 2, 3, or 4 radiographic severity, as defined by the modified Kellgren-Lawrence classification

Exclusion Criteria:

* Pregnant or lactating women
* Women of childbearing potential unwilling to use two forms of contraception
* Cognitively impaired adults.
* Presence of large meniscal tears ("bucket handle" tears), as detected by clinical examination or by magnetic resonance imaging.
* Inflammatory or postinfectious arthritis.
* More than 5 degrees of varus or valgus deformity.
* Kellgren Lawrence grade 4 osteoarthritis in two compartments (the medial or lateral compartments of the tibiofemoral joint or the patellofemoral compartment) in persons over 60 years of age.
* Intraarticular corticosteroid injection within the previous 3 months.
* A major neurologic deficit.
* Serious medical illness with a life expectancy of less than 1 year.
* Prior admission for substance abuse
* Body Mass Index (BMI) of 40 kg/m2 or greater
* Patient receiving experimental medication or participating in another clinical study within 30 days of signing the informed consent
* In the opinion of the investigator or the sponsor the patient is unsuitable for cellular therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2018-11 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 3 months and 12 months

SECONDARY OUTCOMES:
Number of participants with a change in joint function from baseline WOMAC assessment | 3 months and 12 months
Number of participants with a change in radiogrpahic evidence of knee OA from baseline Kellegren-Lawrence grading system | 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Salomon Dayan, MD, Principal Investigator
Locations (1):
- Stem Cell Instsitute, Panama City, Panama